CLINICAL TRIAL: NCT07329465
Title: Comparative Effects of Tabata Training and Periodized Resistance Training on Power, Speed and Agility in Sprinters.
Brief Title: Comparative Effects of Tabata Training and Periodized Resistance Training in Sprinters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0474
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Tabata Training; Periodized Resistance Training; Sprinters

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Group A were receiving periodized resistance training program started with warm up and continued by some exercises such as smith press, seated press, squat, lying dumbbell leg cruel, leg press, lying burble extension, sit up and finally the subjects cooled down.
  Interventions: Other: Periodized Resistance Training
- Group B (Other): Group B were receiving Tabata protocol began with participants performing thrusters as fast as possible for 20 seconds, followed by 10 seconds of resting. The cycle was repeated 7 times for a total of 8 repetitions in 4 minutes.
  Interventions: Other: Tabata Training

INTERVENTIONS:
Other: Periodized Resistance Training — Group A were receiving periodized resistance training program started with warm up and continued by some exercises such as smith press, seated press, squat, lying dumbbell leg cruel, leg press, lying burble extension, sit up and finally the subjects cooled down. At the beginning of the study, the exercises was conducted, 60% intensity while eight maximum repetition and 10% intensity were be added after every two weeks.
  Arms: Group A
Other: Tabata Training — Group B were receiving Tabata training.the Tabata protocol began with participants performing thrusters as fast as possible for 20 seconds, followed by 10 seconds of resting. During the active part, participants will be encouraged to reach near 100% of their HR max. The cycle was repeated 7 times for a total of 8 repetitions in 4 minutes. After completing the protocol, a 5-minute cool-down period (slow walking and stretching exercises) was completed
  Arms: Group B

SUMMARY:
This was a parallel group randomized control trail that utilized purposive sampling to recruit 32 participants. The 32 students are divided into 2 groups, namely the group of Tabata Training and Periodized Resistance Training. Periodized resistance training exercises will be performed three days a week during the eight-week period in group A. The periodized resistance training program started with warm up and continued by some exercises such as smith press, seated press, squat, lying dumbbell leg cruel, leg press, lying burble extension, sit up and finally the subjects cooled down. At the beginning of the study, the exercises will be conducted 60% intensity while eight maximum repetition and 10% intensity will be added after every week. The cycle will be repeated 1 times each exercise for a total of 8 repetitions. Each exercise will performed individually by each participant in a group activity. Tabata training will be performed in group B that included their Exercise sessions started with a general warm-up, and then stretching session followed by a specific warmup. The general warm-up consisted of 5 minutes of marching in place at 60% of the estimated maximal heart rate (HR max= 220 - age) measured with a heart rate monitor. The stretching session included major muscle groups and joints including triceps, deltoid, trapezius, neck extensors, pectoralis, biceps, latissimus dorsi, hamstrings, quadriceps, and gastrocnemius. Each stretch will maintained for 15 to 20 seconds. Then, a specific warm-up session followed that included 2 thruster repetitions of 30 seconds each, followed by 30 seconds of rest. Thrusters are a combination of 2 strength-training exercises: squat and overhead press. After the specific warm-up will be completed, the Tabata protocol began with participants performing thrusters as fast as possible for 20 seconds, followed by 10 seconds of resting. During the active part, participants will encouraged to reach near 100% of their HR max. Intensity will evaluated with heart rate monitors and also with the Borg rating of perceived exertion. The cycle will be repeated 7 times for a total of 8 repetitions in 4 minutes. After completing the protocol, a 5-minute cool-down period (slow walking and stretching exercises) was completed. Total duration of the Tab protocol will be approximately 19 to 20 minutes and will be completed 3 times per week for 8 consecutive weeks

DETAILED DESCRIPTION:
It will be a randomized clinical trial study. The sample size of study will be 38 participants (19 in each group) through non-probability purposive sampling technique. Data will be collected from Pakistan sports board coaching center, model town club Lahore, Sport complex phase 5 sector G DHA Lahore. Data will be collected within 10 months after approval of synopsis.

Inclusion Criteria:

Age group between 18 to 35year. Both male and female of sprinter athletes. Athletes currently performing Regular Training. 100m Sprinters. (should be registered Last 12 months.) [11] Shoe wear (heel drop minimum 1 inch and weight about 150g). [12]

Exclusion Criteria:

Athletes currently perform high resistance training. Injury report half a year ago. Non-sprinting populations. [13] Cardiac and metabolic disorder. Any diagnosed psychological condition that could affect participation. [14] The participants having any supplements or anabolic steroids that could effect performance.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 to 35year.
* Both male and female of sprinter athletes.
* Athletes currently performing Regular Training.
* 100m Sprinters. (should be registered Last 12 months.) [11]
* Shoe wear (heel drop minimum 1 inch and weight about 150g).

Exclusion Criteria:

* Athletes currently perform high resistance training.
* Injury report half a year ago.
* Non-sprinting populations. [13]
* Cardiac and metabolic disorder.
* Any diagnosed psychological condition that could affect participation. [14]
* The participants having any supplements or anabolic steroids that could effect performance.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
30m sprint test | 8 weeks
  The 30m sprint test is used to measure an athlete's acceleration, maximum speed, and speed endurance, assessing their overall sprint power and effectiveness for sports.
Agility T test | 8 weeks
  The Agility T-test is commonly used to assess the ability of team sport athletes to change direction, including acceleration, deceleration, and lateral movement during preseason testing protocols
Vertical Jump Test | 8 weeks
  A vertical jump test measures lower body explosive power by calculating the difference between your standing reach and the highest point you can touch in a jump, often using a wall with chalk or specialized equipment to assess athletic ability for sports

CONTACTS AND LOCATIONS:
Overall Officials: Amina Amjad, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colyer SL, Nagahara R, Takai Y, Salo AIT. How sprinters accelerate beyond the velocity plateau of soccer players: Waveform analysis of ground reaction forces. Scand J Med Sci Sports. 2018 Dec;28(12):2527-2535. doi: 10.1111/sms.13302. Epub 2018 Oct 10. PMID 30230037
- [Background] Haugen T, Seiler S, Sandbakk O, Tonnessen E. The Training and Development of Elite Sprint Performance: an Integration of Scientific and Best Practice Literature. Sports Med Open. 2019 Nov 21;5(1):44. doi: 10.1186/s40798-019-0221-0. PMID 31754845
- [Background] Haugen TA, Breitschadel F, Seiler S. Sprint mechanical variables in elite athletes: Are force-velocity profiles sport specific or individual? PLoS One. 2019 Jul 24;14(7):e0215551. doi: 10.1371/journal.pone.0215551. eCollection 2019. PMID 31339890
- [Background] Healy R, Kenny IC, Harrison AJ. Resistance Training Practices of Sprint Coaches. J Strength Cond Res. 2021 Jul 1;35(7):1939-1948. doi: 10.1519/JSC.0000000000002992. PMID 30747902
- [Background] Haugen T, McGhie D, Ettema G. Sprint running: from fundamental mechanics to practice-a review. Eur J Appl Physiol. 2019 Jun;119(6):1273-1287. doi: 10.1007/s00421-019-04139-0. Epub 2019 Apr 8. PMID 30963240